CLINICAL TRIAL: NCT04477499
Title: Ablation of Ventricular Tachycardia Guided by Multi-site Pacing Using Parallel Mapping
Brief Title: Parallel Mapping for Ventricular Tachycardia
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Jakub Sroubek, Principal Investigator, The Cleveland Clinic
Other Study IDs: IRB 20-470
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Ventricular Tachycardia (V-Tach); Implantable Cardioverter Defibrillator (ICD); Arrythmia
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Catheter ablation in patients with ventricular tachycardia using a new mapping algorithm called, parallel mapping, that is aimed to increase the specificity of mapping and the outcome of ablation.

DETAILED DESCRIPTION:
In patients with scar in the hearts after heart attacks, the risk for dangerous abnormal heart rhythms, including sudden death is high. This is because dead muscle fibers are replaced by scar tissue, creating a physiological condition promoting abnormal heart rhythms.These abnormal heart rhythms are called ventricular arrhythmias or ventricular tachycardias. In these patients, ablation procedures can be helpful, however the recurrence rate of arrhythmias after ablation remains unacceptably high. The primary reason for this high recurrence rate is nonspecific mapping methodologies for identifying the heart area responsible for these arrhythmias. Therefore, new methods for increasing the specificity of mapping have been the subject of significant research for many years, however implementation of these methods in clinical practice has been challenged by limited technologies. Recently, a new mapping technology named "parallel mapping" has been developed, received FDA approval and is routinely utilized at the Cleveland Clinic. However, the workflow of using parallel mapping, and the efficacy of ablation using this technology have not been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* History of scar-mediated sustained ventricular tachycardia
* Failure of therapy with Anti arrhythmic drugs
* Implanted ICD or a plan for ICD implantation after the ablation
* Willingness to adhere to the study restrictions and comply with all post procedural follow-up requirements
* Ability to understand the requirements of the study and sign an informed consent

Exclusion Criteria:

* Patients with reversible causes of ventricular tachycardia including ongoing ischemia or electrolyte abnormalities
* Contraindication to anticoagulation therapy
* Stroke within 30 days before enrollment
* Life expectancy <1 year
* Individual has a known, unresolved history of drug use or alcohol dependency lacks the ability to comprehend or follow instructions or would be unlikely or unable to comply with study follow-up requirements
* Pregnant or breast feeding at time of signing consent
* Patient undergoing cardiac transplantation
* Enrolled or participates in other drug or device studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with history of scar-mediated recurrent ventricular tachycardia, who had failed therapy with anti arrhythmic drugs. All patients are planned to undergo catheter ablation procedure for ventricular tachycardia as part of the usual clinical care. All patients who meet the eligibility criteria may be included in the study regardless of gender, race or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Single procedure freedom from ventricular recurrence at 1 year | 12 months
  Number of VT

SECONDARY OUTCOMES:
Freedom from implantable cardioverter defibrillator (ICD) shocks | 12 months
  Number of ICD shocks
Reduction in mapping time using parallel mapping algorithm | 12 months
  Minutes
Reduction in radiofrequency ablation time | 12 months
  Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Sroubek, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No